CLINICAL TRIAL: NCT07144449
Title: Effect of Information-based Symptom Management on the Quality of Life of Cancer Patients
Brief Title: Nurse-Led Electronic Patient-Reported Outcome System to Improve Quality of Life in Chemotherapy Patients
Acronym: NURSE-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHIAO-CHI KUAN (Other)
Responsible Party: Sponsor-Investigator, CHIAO-CHI KUAN, Registered Nurse (RN), National Taiwan University
Organization: National Taiwan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202304084RIND; NTUCCS-112-23 (Other Grant/Funding Number: National Taiwan University Cancer Center, NTUCC)
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Neoplasms; Nursing Caries
Keywords: oncology; nurse care; digital health
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the intervention group (nurse-led ePRO system) or control group (usual care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nurse-Led ePRO System (Experimental): Participants will use a nurse-led electronic patient-reported outcome (ePRO) system during chemotherapy. The system was designed by oncology nurses and allows patients to complete weekly symptom assessments for 12 weeks. Automated feedback and evidence-based self-care advice are provided. Alerts are triggered for severe symptoms, prompting follow-up by oncology nurses including weekly phone calls.
  Interventions: Behavioral: Nurse-Led ePRO System
- Usual Care (Active Comparator): Participants will receive standard oncology care without access to the ePRO system. Symptom monitoring and management will be provided according to routine clinical practice by the treating oncology team.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Nurse-Led ePRO System — A nurse-designed electronic patient-reported outcome (ePRO) system for chemotherapy patients. Participants complete weekly symptom assessments for 12 weeks through an electronic platform. The system provides automated feedback, evidence-based self-care advice, and alerts to oncology nurses. Nurses follow up with weekly phone calls if severe symptoms are reported. This intervention is intended to improve symptom self-management, quality of life, and health literacy.
  Arms: Nurse-Led ePRO System
Behavioral: Usual Care — Participants will receive standard oncology care without the use of an ePRO system. Symptom monitoring and management will be provided according to routine clinical practice by the treating oncology team, typically during scheduled visits or when patients proactively report problems.
  Arms: Usual Care

SUMMARY:
Chemotherapy often causes burdensome symptoms that affect daily life and reduce patients' quality of life. This study aims to test whether an information-based symptom management program can help cancer patients better manage their symptoms, improve self-care ability, and enhance quality of life. The program was developed by nurses and delivered through a simple electronic platform, allowing patients to report symptoms such as fever, pain, shortness of breath, nausea, diarrhea, fatigue, or anxiety. Patients in the intervention group will receive tailored self-care advice and weekly nurse follow-up calls, while the control group will receive usual care. The study will compare outcomes in symptom self-management, quality of life, and health literacy between the two groups over 12 weeks.

DETAILED DESCRIPTION:
This study is a single-center, two-arm, parallel-group randomized controlled trial designed to evaluate the effectiveness of a nurse-led electronic patient-reported outcome (ePRO) system for symptom management in patients receiving chemotherapy. Participants will be randomized 1:1 into the intervention group or control group.

Intervention group: Participants will use the nurse-led ePRO system to report weekly symptoms over 12 weeks. The system automatically provides tailored, evidence-based self-care advice and triggers nurse follow-up, including weekly phone calls when severe symptoms are reported.Control group: Participants will receive standard oncology care without access to the ePRO system. Symptom monitoring and management will follow routine clinical practice.Three validated tools will be used to measure outcomes at four time points (baseline, week 4, week 8, and week 12):

Partners in Health (PIH) Scale - symptom self-management Functional Assessment of Cancer Therapy-General (FACT-G) - quality of life Mandarin Multidimensional Health Literacy Questionnaire (MMHLQ) - health literacy

The primary outcomes are changes in self-management and quality of life, while the secondary outcome is health literacy. Statistical analyses will follow the intention-to-treat principle, and group differences over time will be evaluated using linear mixed-effects models.

This trial aims to provide high-quality evidence on the effectiveness of a nurse-led, digitally delivered intervention for improving self-management, quality of life, and health literacy in patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

- Adults aged 18 years or older

Diagnosis of cancer and currently receiving chemotherapy

Able to communicate in Mandarin Chinese

Access to and ability to use a smartphone or tablet with internet connection

Provide written informed consent

Exclusion Criteria:

Cognitive impairment, severe psychiatric illness, or any condition that limits ability to complete questionnaires

Physical or medical conditions judged by the treating physician to interfere with study participation

Participation in another interventional trial that could confound study outcomes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-05-04 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life | Baseline, Week 4, Week 8, Week 12
  Quality of life will be assessed using the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire. The FACT-G contains 27 items across four domains: Physical, Social/Family, Emotional, and Functional well-being. The total score ranges from 0 to 108, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Self-Management | Baseline, Week 4, Week 8, Week 12
  Symptom self-management will be evaluated using the Partners in Health (PIH) Scale. The PIH consists of 12 items scored on a 9-point Likert scale. The total score ranges from 0 to 96, with higher scores indicating better self-management ability.
Health Literacy | Baseline, Week 4, Week 8, Week 12
  The MMHLQ includes 20 items rated on a 4-point Likert scale. The total score ranges from 20 to 80, with higher scores indicating better health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Hsueh-Hsing Pan, RN, PhD, Principal Investigator — Graduate Institute of Nursing, School of Nursing, National Defense Medical Center, Taipei, Taiwan
Locations (1):
- National Taiwan University Cancer Center, Taipei County, Taipei, Taiwan